CLINICAL TRIAL: NCT07029997
Title: Post-Market Clinical Follow-Up Study of the Solo+ Tympanostomy Tube Device
Status: Not yet recruiting | Type: Observational
Sponsor: AventaMed DAC (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP004
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Otitis Media; Middle Ear Infections
Keywords: ear tubes
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adults and pedriatic patients who have had eartubes inserted, both prospective and retrospective.
  Interventions: Device: Solo+ Tympanostomy Tube Device (Solo+ TTD)

INTERVENTIONS:
Device: Solo+ Tympanostomy Tube Device (Solo+ TTD) — insertion of eartubes

SUMMARY:
The purpose of this project is to collect information from the doctor notes about the use of the device, to monitor the tubes after surgery, and collect information from patients and parents/guardians about their views on the procedure. Since the device became available in Europe, it is important to collect information from both patients planned for the procedure (prospective) and those who already underwent the procedure (retrospective) to have collect as much data as possible.

DETAILED DESCRIPTION:
Patients are being asked to participate in this study because they have been treated, will be treated, or have undergone a treatment attempt with the Solo+ Tympanostomy Tube Device (Solo+ TTD), manufactured by AventaMed. The Solo+ TTD device is a CE marked device designed to deploy ear tubes across the ear drum.

Ear tubes (also known as tympanostomy tubes or ventilation tubes) are predominantly used in treating repeated or long-term middle ear infections, or to treat a build-up of fluid in the middle ear, mostly in children, yet also used for adults. Ear tube insertion allows for air to ventilate the middle ear space and drain fluid from the middle ear.

The Solo+ Tympanostomy Tube Device (Solo+ TTD) is an all-in-one device for the insertion of ear tubes using as little as topical anaesthesia, without requiring general anaesthesia as is the case for other similar devices. The Solo+ TTD is approved for use in children and adults. It is available in Europe and already in use by some clinics and hospitals.

The purpose of this study is to collect information about the use the Solo+ TTD.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or Parent/Guardian is able to understand the information document and (depending in the country's legislation) does not object participating or is willing to provide documented informed consent
* Subject was or will be treated, or had a treatment attempted with the study device.

Exclusion Criteria:

* None

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and paediatric patients (over 6 months) requiring tympanostomy tube placement treated with Solo+ TTD. It is anticipated at least 75% of the study population will be comprised of paediatric patients (under 18 years of age)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Procedure Success (Performance) | 48 months
  Percentage of subjects in which the tympanostomy tube is inserted in all indicated ears in a single procedure without the need to schedule a secondary procedure
Functioning Tubes (Performance) | 48 months
  Percentage of ears with a functioning tube (without extrusion and without occlusion) at standard of care follow-up visits until tube extrusion or discharge from standard clinical care
Early Adverse Event (AE) Rates (Safety) | 48 months
  Incidence and nature of device- or procedure-related AEs (per ear and per subject) from the day of the procedure to first follow-up visit post procedure